CLINICAL TRIAL: NCT06422143
Title: Phase 3 Study of Pembrolizumab in Combination With Carboplatin/Taxane (Paclitaxel or Nab-paclitaxel) Followed by Pembrolizumab With or Without Maintenance MK-2870 in the First-line Treatment of Metastatic Squamous Non-small Cell Lung Cancer
Brief Title: Pembrolizumab With or Without Maintenance Sacituzumab Tirumotecan (Sac-TMT; MK-2870) in Metastatic Squamous Non-small Cell Lung Cancer (NSCLC) [MK-2870-023]
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2870-023; 2023-510128-66-00 (Registry Identifier: EU CT); U1111-1301-2790 (Registry Identifier: UTN); jRCT2021240015 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); MK-2870-023 (Other: MSD)
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Participants are allocated to a single induction arm, then assigned randomly to one of 2 maintenance arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maintenance Arm A: Pembrolizumab + sac-TMT (Experimental): During the Induction phase, participants receive pembrolizumab 200 mg q3w for 4 cycles, carboplatin area under the curve (AUC) 6 (mg/mL/min) q3w for 4 cycles, and paclitaxel 200 mg/m2 q3w for 4 cycles or nab-paclitaxel 100 mg/m2 weekly for 4 cycles. Note: per investigator discretion, carboplatin AUC 5 mg/mL/min q3w or paclitaxel 175mg/m2 q3w may be administered.
  During the Maintenance phase, participants receive sac-TMT 4 mg/kg infusion every 2 weeks (q2w) until discontinuation criteria is met for sac-TMT; and pembrolizumab 400 mg every 6 weeks (q6w) for 96 weeks.
  Interventions: Biological: Pembrolizumab; Biological: sac-TMT; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel
- Maintenance Arm B: Pembrolizumab Monotherapy (Active Comparator): During the Induction phase, participants receive pembrolizumab 200 mg q3w for 4 cycles, carboplatin AUC 6 (mg/mL/min) q3w for 4 cycles, and paclitaxel 200 mg/m2 q3w for 4 cycles or nab-paclitaxel 100 mg/m2 weekly for 4 cycles.
  During the Maintenance phase, participants receive pembrolizumab 400 mg q6w for 96 weeks.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel

INTERVENTIONS:
Biological: Pembrolizumab — Intravenous (IV) infusion
  Other Names: KEYTRUDA®; MK-3475; SCH 900475
Biological: sac-TMT — IV infusion
  Other Names: MK-2870; Sacituzumab tirumotecan
  Arms: Maintenance Arm A: Pembrolizumab + sac-TMT
Drug: Carboplatin — Participants receive AUC 6 or AUC 5 mg/mL/min IV infusion on Day 1 of each 21-day cycle for 4 cycles as background therapy during the study.
Drug: Paclitaxel — Participants receive 200 mg/m^2 or 175 mg/m^2 IV infusion on Day 1 of each 21-day cycle for 4 cycles as background therapy during the study.
Drug: Nab-paclitaxel — Participants receive 100 mg/m^2 IV infusion on Days 1, 8 and 15 of each 21-day cycle for 4 cycles as background therapy during the study.

SUMMARY:
This is a phase 3 study of pembrolizumab in combination with carboplatin/taxane (paclitaxel or nab-paclitaxel) followed by pembrolizumab with or without maintenance sacituzumab tirumotecan (sac-TMT; MK-2870) in first-line treatment of metastatic squamous non-small cell lung cancer. It is hypothesized that pembrolizumab with maintenance sacituzumab tirumotecan is superior to pembrolizumab without sacituzumab tirumotecan maintenance with respect to overall survival (OS).

DETAILED DESCRIPTION:
All participants undergo an initial induction phase of four cycles, each cycle consisting of pembrolizumab q3w + carboplatin q3w + paclitaxel q3w or nabpaclitaxel weekly. Participants are then randomly assigned to pembrolizumab maintenance vs. pembrolizumab + sac-TMT maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of squamous non-small cell lung cancer (NSCLC) [Stage IV: M1a, M1b, M1c, American Joint Committee on Cancer Staging Manual, version 8]
* Measurable disease per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 as assessed by the local site investigator/radiology
* Has life expectancy ≥3 months
* Has Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1 assessed within 7 days prior to allocation
* Archival tumor tissue sample or newly obtained core, incisional, or excisional biopsy of a tumor lesion not previously irradiated has been provided
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART)
* Participants who are hepatitis B surface antigen (HBsAg)-positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load before allocation
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening
* Participants who have adverse events (AEs) due to previous anticancer therapies must have recovered to Grade ≤1 or baseline (participants with endocrine-related AEs who are adequately treated with hormone replacement are eligible)
* Has adequate organ function
* For Maintenance only (prior to randomization): is without disease progression of their NSCLC, as determined by BICR using RECIST 1.1 after completion of study-specified Induction with an evaluable scan at Week 12 or most recent scan before randomization
* For Maintenance only (prior to randomization): has ECOG PS of 0 or 1 as assessed at the Prerandomization Visit
* For Maintenance only (prior to randomization): all AEs (with the exception of alopecia, Grade ≤2 fatigue, Grade ≤2 peripheral neuropathy, and Grade ≤2 endocrine-related AEs requiring treatment or hormone replacement) have recovered

Exclusion Criteria:

* Diagnosis of small cell lung cancer or, for mixed tumors, presence of small cell elements
* History of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing
* Active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea)
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, uncontrolled symptomatic arrhythmia, prolongation of QTcF interval to >480 ms, and other serious cardiovascular and cerebrovascular diseases within 6 months before study intervention
* HIV-infected participants who have been newly diagnosed or with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Received prior systemic chemotherapy or other targeted or biological antineoplastic therapy for their metastatic NSCLC. Note: Prior treatment with chemotherapy and/or radiation as a part of neoadjuvant or adjuvant therapy or chemoradiation therapy for nonmetastatic NSCLC is allowed as long as therapy was completed at least 12 months before diagnosis of metastatic NSCLC
* Received prior therapy with an anti-programmed cell death 1 protein (PD-1), anti-programmed cell death ligand 1 (PD-L1), or anti programmed cell death ligand 2 (PD-L2) agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, cytotoxic T lymphocyte-associated protein 4, OX-40, CD137). Note: Prior treatment with an anti-PD-1 or anti-PD-L1 agent for nonmetastatic NSCLC is allowed as long as therapy was completed at least 12 months before diagnosis of metastatic NSCLC
* Received prior treatment with a trophoblast cell-surface antigen 2 (TROP2)-targeted antidrug conjugate (ADC)
* Received radiation therapy to the lung that is >30 Gray within 6 months of start of study intervention
* Received prior radiotherapy within 2 weeks of start of study intervention, or radiation-related toxicities, requiring corticosteroids
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Participants who have not adequately recovered from major surgery or have ongoing surgical complications
* Received prior treatment with a topoisomerase I inhibitor-containing ADC
* Is currently receiving a strong inducer/inhibitor of CYP3A4 that cannot be discontinued for the duration of the study (the required washout period before starting sac-TMT is 2 weeks)
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has known central nervous system (CNS) metastases/carcinomatous meningitis
* Severe hypersensitivity (≥Grade 3) to study intervention and/or any of its excipients or to another biologic therapy
* Active autoimmune disease that has required systemic treatment in the past 2 years (replacement therapy [eg, thyroxine, insulin, or physiologic corticosteroid] is allowed)
* History of (noninfectious)pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Active infection requiring systemic therapy
* History of allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 851 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2029-01-12 (Estimated); Study Completion 2031-02-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to ~50 months
  OS is the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to ~79 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Number of Participants With ≥1 Adverse Event (AE) | Up to ~79 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Discontinuing from Study Therapy Due to AE(s) | Up to ~79 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Change in Score from Baseline to a Predefined Timepoint in Participant-Reported Global health status/Quality of Life (QoL) Score (EORTC QLQ-C30 Items 29 and 30) | Baseline and up to ~79 months
  European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) is a 30-item scale to assess the overall quality of life in cancer patients. The global health status and QoL scores are based on participant responses to items 29 ("How would you rate your overall health during past week?") and 30 ("How would you rate your overall quality of life during the week?") that are scored on a 7-point scale (1 = "Very poor" to 7 = "Excellent"). Higher scores indicate better overall health status.
Change in Score from Baseline to a Predefined Timepoint in Participant-Reported Dyspnea (EORTC QLQ-C30 Item 8) | Baseline and up to ~79 months
  EORTC QLQ-C30 is a 30-item scale to assess the overall quality of life of cancer patients. The dyspnea score is based on participant responses to item 8 ("Were you short of breath?") that is scored on a 4-point scale (1 = 'Not at All' to 4 = 'Very Much'). Higher scores indicate worse dyspnea symptoms.
Change in Score from Baseline to a Predefined Timepoint in Participant-Reported Cough (EORTC QLQ-LC13 Item 31) | Baseline and up to ~79 months
  EORTC QLQ-C13 is a 13-item addendum to EORTC QLQ-C30 to assess the overall quality of life of lung cancer patients. The cough score is based on participant responses to item 31 ("How much did you cough?") that is scored on a 4-point scale (1 = 'Not at All' to 4 = 'Very Much'). Higher scores indicate worse cough.
Change in Score from Baseline to a Predefined Timepoint in Participant-Reported Chest Pain (EORTC QLQ-LC13 Item 40) | Baseline and up to ~79 months
  EORTC QLQ-C13 is a 13-item addendum to EORTC QLQ-C30 to assess the overall quality of life of lung cancer patients. The chest pain score is based on participant responses to item 40 e (1 = "Not at All" to 4 = "Very Much").
Time to First Deterioration (TTD) in Global Health Status/QoL Scores (EORTC QLQ-C30 Items 29 and 30) | Up to ~79 months
  EORTC QLQ-C30 is a 30-item scale to assess the overall quality of life in cancer patients. TTD in global health status and QoL scores are based on participant responses to items 29 ("How would you rate your overall health during past week?") and 30 ("How would you rate your overall quality of life during the week?") that are scored on a 7-point scale (1 = "Very poor" to 7 = "Excellent"). Higher scores indicate better overall health status.
TTD in Dyspnea Score (EORTC QLQ-C30 Item 8) | Up to ~79 months
  EORTC QLQ-C30 is a 30-item scale to assess the overall quality of life of cancer patients. TTD in dyspnea score is based on participant responses to item 8 ("Were you short of breath?") that is scored on a 4-point scale (1 = 'Not at All' to 4 = 'Very Much'). Higher scores indicate worse dyspnea symptoms.
TTD in Cough Score (EORTC QLQ-LC13 Item 31) | Up to ~79 months
  EORTC QLQ-C13 is a 13-item addendum to EORTC QLQ-C30 to assess the overall quality of life of lung cancer patients. TTD in cough score is based on participant responses to item 31 ("How much did you cough?") that is scored on a 4-point scale (1 = 'Not at All' to 4 = 'Very Much'). Higher scores indicate worse cough.
TTD in Chest Pain Score (EORTC QLQ-LC13 Item 40) | Up to ~79 months
  EORTC QLQ-C13 is a 13-item addendum to EORTC QLQ-C30 to assess the overall quality of life of lung cancer patients. TTD in chest pain score is based on participant responses to item 40 ("Have you had pain in your chest?") that is scored on a 4-point scale (1 = 'Not at All' to 4 = 'Very Much'). Higher scores indicate worse chest pain.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (203):
- United States (17):
  - CARTI Cancer Center ( Site 0006), Little Rock, Arkansas
  - Roy and Patricia Disney Family Cancer Center - Providence Saint Joseph Medical Center ( Site 0122), Burbank, California
  - Exempla Lutheran Medical Center ( Site 0119), Golden, Colorado
  - Intermountain Health St. Mary's Regional Hospital ( Site 0116), Grand Junction, Colorado
  - Mid Florida Hematology and Oncology Center ( Site 0109), Orange City, Florida
  - Centricity Research Columbus Cancer Center ( Site 0111), Columbus, Georgia
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital ( Site 0001), Marietta, Georgia
  - Southeastern Regional Medical Center ( Site 0004), Newnan, Georgia
  - University of Chicago Medical Center ( Site 0145), Chicago, Illinois
  - Allina Health Cancer Institute - Abbott Northwestern Hospital ( Site 0146), Minneapolis, Minnesota
  - New Mexico Oncology Hematology Consultants Ltd. ( Site 0123), Albuquerque, New Mexico
  - University of New Mexico Comprehensive Cancer Center ( Site 0135), Albuquerque, New Mexico
  - St Luke's University Health Network ( Site 0017), Bethlehem, Pennsylvania
  - Thomas Jefferson University - Clinical Research Institute ( Site 0147), Philadelphia, Pennsylvania
  - Memorial Hermann Cancer Center ( Site 0015), Houston, Texas
  - Oncology Consultants P.A. ( Site 0124), Houston, Texas
  - Mays Cancer Center ( Site 0132), San Antonio, Texas
- Argentina (6):
  - Instituto Alexander Fleming ( Site 0203), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0200), Mar del Plata, Buenos Aires
  - Instituto Médico Río Cuarto ( Site 0204), Río Cuarto, Córdoba Province
  - Fundacion Intecnus ( Site 0205), Bariloche, Río Negro Province
  - Sanatorio Parque ( Site 0201), Rosario, Santa Fe Province
  - Hospital Aleman-Oncology ( Site 0202), Buenos Aires
- Austria (4):
  - Ordensklinikum Linz GmbH Elisabethinen-Department of Pneumology ( Site 0720), Linz, Upper Austria
  - Klinik Hietzing ( Site 0740), Vienna
  - Standort Penzing der Klinik Ottakring-Abteilung für Atemwegs-und Lungenkrankheiten ( Site 0730), Vienna
  - Klinik Floridsdorf-Abteilung für Innere Medizin und Pneumologie ( Site 0710), Vienna
- Brazil (7):
  - Hospital do Cancer de Pernambuco ( Site 0312), Recife, Pernambuco
  - Vencer Centro de Pesquisa Clínica ( Site 0309), Teresina, Piauí
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre ( Site 0311), Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição ( Site 0300), Porto Alegre, Rio Grande do Sul
  - Instituto de Oncologia Saint Gallen ( Site 0304), Santa Cruz do Sul, Rio Grande do Sul
  - Hospital de Base de São José do Rio Preto ( Site 0310), São José do Rio Preto, São Paulo
  - Hospital Paulistano ( Site 0307), São Paulo
- Canada (5):
  - Kingston Health Sciences Centre-Kingston General Hospital Site ( Site 0100), Kingston, Ontario
  - Waterloo Regional Health Network (WRHN) ( Site 0153), Kitchener, Ontario
  - St. Marys Hospital Center ( Site 0105), Montreal, Quebec
  - McGill University Health Centre ( Site 0103), Montreal, Quebec
  - Centre integre universitaire de sante et de services sociaux de la Mauricie-et-du-centre-du-quebec ( Site 0106), Trois-Rivières, Quebec
- Chile (6):
  - Centro de Investigación del Maule ( Site 0419), Talca, Maule Region
  - FALP ( Site 0409), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-Hemato-Oncology ( Site 0402), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0407), Santiago, Region M. de Santiago
  - ONCOCENTRO APYS-ACEREY ( Site 0400), Viña del Mar, Región de Valparaíso
  - Bradford Hill Norte ( Site 0420), Antofagasta
- China (28):
  - Beijing Cancer Hospital ( Site 2411), Beijing, Beijing Municipality
  - Beijing Cancer hospital-intrathoratic deparmtment II ( Site 2410), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 2412), Beijing, Beijing Municipality
  - Army Medical Center of People's Liberation Army-respiratory ( Site 2426), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 2419), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University-oncology ( Site 2420), Xiamen, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University ( Site 2417), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital-Depatrment of Respiratory and Critical Care Medicine ( Site 2416), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital-oncology of department ( Site 2415), Harbin, Heilongjiang
  - Henan Cancer Hospital-Pneumology department ( Site 2423), Zhengzhou, Henan
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 2424), Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University-Oncology ( Site 2418), Changsha, Hunan
  - First Huai'an Hospital Affiliated to Nanjing Medical University ( Site 2402), Huai'an, Jiangsu
  - Northern Jiangsu People's Hospital-General Surgery Department ( Site 2403), Yangzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University-Oncology Department ( Site 2405), Nanchang, Jiangxi
  - The First affiliated hospital of Nanchang University (Xianghu campus) ( Site 2404), Nanchang, Jiangxi
  - Jilin Province Tumor Hospital-GCP office ( Site 2413), Changchun, Jilin
  - The First Hospital of Jilin University-Oncology ( Site 2414), Changchun, Jilin
  - Shanghai East Hospital ( Site 2428), Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital ( Site 2427), Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University ( Site 2422), Chengdu, Sichuan
  - Sichuan Cancer hospital. ( Site 2421), Chengdu, Sichuan
  - The Affiliated Cancer Hospital of Xinjiang Medical University ( Site 2425), Ürümqi, Xinjiang
  - The first Affiliated Hospital, Zhejiang University School of Medicine-Respiratory Department ( Site 2406), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine-Medical Oncology ( Site 2407), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital-Breast Oncology ( Site 2408), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province ( Site 2430), Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University-Respiratory department ( Site 2409), Wenzhou, Zhejiang
- Colombia (5):
  - Centro Cancerológico del Caribe (CECAC) ( Site 0509), Barranquilla, Atlántico
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 0500), Bogotá, Bogota D.C.
  - Sociedad De Oncología y Hematología Del Cesar SAS-Oncology ( Site 0501), Valledupar, Cesar Department
  - Oncologos del Occidente ( Site 0504), Pereira, Risaralda Department
  - Fundación Valle del Lili-Oncology CIC ( Site 0505), Cali, Valle del Cauca Department
- Czechia (4):
  - Masarykuv onkologicky ustav-Klinika komplexni onkologicke pece ( Site 0800), Brno, Brno-mesto
  - Nemocnice AGEL Ostrava - Vitkovice a.s.-Plicni oddeleni ( Site 0803), Ostrava-Vitkovice, Ostrava Mesto
  - Multiscan-Onkologicke a radiologicke centrum Multiscan Pardubice ( Site 0804), Pardubice, Pardubický kraj
  - Fakultni nemocnice Olomouc-Klinika plicnich nemoci a tuberkulozy ( Site 0802), Olomouc
- France (6):
  - Clinique Clairval ( Site 0904), Marseille, Bouches-du-Rhone
  - Hôpital Robert Schuman ( Site 0907), Vantoux, Lorraine
  - Institut de Cancérologie de l'Ouest ( Site 0908), Angers, Maine-et-Loire
  - Sainte Catherine Institut du Cancer Avignon Provence ( Site 0902), Avignon, Vaucluse
  - CHD Vendee ( Site 0901), La Roche-sur-Yon, Vendee
  - Hôpital Saint-Louis ( Site 0906), Paris
- Germany (5):
  - GEFOS Gesellschaft f. onkologische Studien ( Site 1005), Dortmund, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung ( Site 1001), Essen, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein-Pneumologie ( Site 1000), Lübeck, Schleswig-Holstein
  - SRH Wald-Klinikum Gera-Zentrum für klinische Studien ( Site 1006), Gera, Thuringia
  - Charité Campus Virchow-Klinikum-Department of Infectious Diseases and Pulmonary Medicine ( Site 1003), Berlin
- Hungary (6):
  - Bacs-Kiskun Varmegyei Oktatokorhaz ( Site 1100), Kecskemét, Bács-Kiskun county
  - Petz Aladar Egyetemi Oktato Korhaz ( Site 1101), Győr, Győr-Moson-Sopron
  - Jász-Nagykun-Szolnok Vármegyei Hetényi Géza Kórház-Onkologiai Kozpont ( Site 1103), Szolnok, Jász-Nagykun-Szolnok
  - Reformatus Pulmonologiai Centrum ( Site 1102), Törökbálint, Pest County
  - Zala Megyei Szent Rafael Kórház ( Site 1110), Zalaegerszeg, Zala County
  - Országos Korányi Pulmonológiai Intézet ( Site 1104), Budapest
- St. James's Hospital ( Site 1200), Dublin, Ireland
- Israel (4):
  - Rambam Health Care Campus-Oncology Division ( Site 1302), Haifa
  - Shaare Zedek Medical Center ( Site 1300), Jerusalem
  - Rabin Medical Center ( Site 1303), Petah Tikva
  - Sheba Medical Center ( Site 1301), Ramat Gan
- Italy (11):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-Oncologia clinica sperimentale Toraco-Polmonare ( Site 1401), Napoli, Campania
  - Azienda Ospedaliera S. Giovanni Addolorata-Oncologia Medica ( Site 1409), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1404), Milan, Lombardy
  - Fondazione IRCCS San Gerardo dei Tintori-Oncologia ( Site 1412), Monza, Lombardy
  - Istituto Clinico Humanitas-U.O di Oncologia medica ed Ematologia ( Site 1408), Rozzano, Milano
  - Istituto Nazionale Tumori Regina Elena-Oncologia Medica 2 ( Site 1402), Rome, Roma
  - Azienda Ospedaliera Spedali Civili di Brescia-Oncology ( Site 1414), Brescia
  - Ospedale San Martino ( Site 1407), Genova
  - Fondazione IRCCS Policlinico San Matteo-Oncology ( Site 1410), Pavia
  - Ospedale di Circolo e Fondazione Macchi Varese-Oncology ( Site 1413), Varese
  - Centro Ricerche Cliniche di Verona s.r.l. c/o Policlinico G.B.Rossi ( Site 1415), Verona
- Japan (24):
  - Aichi Cancer Center ( Site 2502), Nagoya, Aichi-ken
  - Nagoya University Hospital ( Site 2519), Nagoya, Aichi-ken
  - Fujita Health University Hospital ( Site 2515), Toyoake, Aichi-ken
  - Hirosaki University Hospital ( Site 2514), Hirosaki, Aomori
  - National Cancer Center Hospital East ( Site 2501), Kashiwa, Chiba
  - Ehime University Hospital ( Site 2511), Tōon, Ehime
  - Gunma Prefectural Cancer Center ( Site 2510), Ōta, Gunma
  - Takarazuka City Hospital ( Site 2508), Takarazuka, Hyōgo
  - Kanazawa University Hospital ( Site 2513), Kanazawa, Ishikawa-ken
  - St. Marianna University Hospital ( Site 2521), Kawasaki, Kanagawa
  - Kanagawa Cardiovascular and Respiratory Center ( Site 2518), Yokohama, Kanagawa
  - Kanagawa Cancer Center ( Site 2504), Yokohama, Kanagawa
  - Matsusaka Municipal Hospital ( Site 2522), Matsusaka, Mie-ken
  - Sendai Kousei Hospital ( Site 2507), Sendai, Miyagi
  - Kansai Medical University Hospital ( Site 2503), Hirakata, Osaka
  - Saitama Prefectural Cancer Center ( Site 2512), Kitaadachi-gun, Saitama
  - Cancer Institute Hospital of JFCR ( Site 2500), Koto, Tokyo
  - Toho University Omori Medical Center ( Site 2520), Ōta-ku, Tokyo
  - National Center for Global Health and Medicine ( Site 2516), Shinjuku, Tokyo
  - National Hospital Organization Yamaguchi Ube Medical Center ( Site 2523), Ube, Yamaguchi
  - Chiba University Hospital ( Site 2517), Chiba
  - National Hospital Organization Kyushu Medical Center ( Site 2509), Fukuoka
  - Niigata Cancer Center Hospital ( Site 2505), Niigata
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute ( Site 2506), Osaka
- Peru (4):
  - Clínica San Antonio ( Site 0606), Trujillo, La Libertad
  - Clínicas AUNA Sede Chiclayo ( Site 0604), Chiclayo, Lambayeque
  - Oncosalud-Clinical Research ( Site 0600), Lima
  - Hospital Militar Central Coronel Luis Arias Schereiber ( Site 0602), Lima
- Poland (9):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 1503), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Regionalny Szpital Specjalistyczny im. dr. Władyslawa Biegańskiego ( Site 1513), Grudziądz, Kuyavian-Pomeranian Voivodeship
  - Szpital Specjalistyczny im. Henryka Klimontowicza ( Site 1507), Gorlice, Lesser Poland Voivodeship
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie-Oncology Department ( Site 1515), Krakow, Lesser Poland Voivodeship
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii-Oddzial Onkologii Klinicznej z Pododdzialem Dz ( Site 1510), Poznań, Lower Silesian Voivodeship
  - Instytut Gruźlicy i Chorób Płuc w Warszawie ( Site 1523), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 1500), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 1501), Przemyśl, Podkarpackie Voivodeship
  - Szpital Wojewódzki w Koszalinie. ( Site 1517), Poland, West Pomeranian Voivodeship
- Romania (8):
  - Centrul Medical Medicover Victoria ( Site 2000), Bucharest, București
  - Cardiomed SRL Cluj-Napoca ( Site 2002), Cluj-Napoca, Cluj
  - SC Radiotherapy Center Cluj SRL-Oncologie Medicala ( Site 2001), Florești, Cluj
  - Centrul de Oncologie Sfantul Nectarie-Medical ( Site 2004), Craiova, Dolj
  - Cabinet Medical Oncomed ( Site 2005), Timișoara, Timiș County
  - SC ONCO CARD SRL ( Site 2007), Brasov
  - Lotus-Med ( Site 2009), Bucharest
  - Clinica Polisano ( Site 2008), Sibiu
- South Korea (8):
  - The Catholic University of Korea, Incheon St. Mary's Hospital ( Site 2106), Bupyeong-gu, Incheon
  - Pusan National University Yangsan Hospital ( Site 2104), Yangsan, Kyongsangnam-do
  - Pusan National University Hospital ( Site 2100), Busan, Pusan-Kwangyokshi
  - Kyungpook National University Chilgok Hospital-Pulmonology ( Site 2102), Deagu, Taegu-Kwangyokshi
  - Chungnam national university hospital-Department of Internal Medicine ( Site 2107), Daejeon, Taejon-Kwangyokshi
  - Kyung Hee University Hospital ( Site 2101), Seoul
  - Asan Medical Center ( Site 2105), Seoul
  - Korea University Guro Hospital-Internal Medicine ( Site 2103), Seoul
- Spain (6):
  - CHUS - Hospital Clinico Universitario-Servicio de Oncologia ( Site 1703), Santiago de Compostela, Galicia
  - Hospital Insular de Gran Canaria-Oncology ( Site 1701), Las Palmas de Gran Canaria, Las Palmas
  - Hospital Quirón Málaga ( Site 1704), Málaga, Malaga
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 1700), Barcelona
  - Hospital Universitario Fundación Jiménez Díaz-Oncology & Hematology ( Site 1702), Madrid
  - Hospital Universitario Virgen de Valme-Departamento de Oncologia ( Site 1705), Seville
- Taiwan (8):
  - National Taiwan University Cancer Center (NTUCC) ( Site 2209), Taipei City, Taipei
  - Taoyuan General Hospital ( Site 2203), Taoyuan, Taoyuan
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 2207), Kaohsiung City
  - Taichung Veterans General Hospital ( Site 2204), Taichung
  - National Cheng Kung University Hospital ( Site 2205), Tainan
  - National Taiwan University Hospital-Oncology ( Site 2208), Taipei
  - Mackay Memorial Hospital-Chest Medicine ( Site 2201), Taipei
  - Chang Gung Medical Foundation-Linkou Branch-Clinic of Chest Medicine ( Site 2202), Taoyuan District
- Thailand (7):
  - Faculty of Medicine Siriraj Hospital ( Site 2301), Bangkok, Bangkok
  - Bangkok Metropolitan Administration Medical College and Vajira Hospital ( Site 2300), Dusit, Bangkok
  - Prapokklao Hospital ( Site 2306), Mueang, Changwat Chanthaburi
  - Faculty of Medicine - Khon Kaen University ( Site 2305), Muang, Changwat Khon Kaen
  - Lampang Cancer Hospital ( Site 2304), Lampang, Changwat Lampang
  - Songklanagarind hospital ( Site 2303), Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital ( Site 2302), Chiang Mai
- Turkey (Türkiye) (8):
  - Medipol Mega Universite Hastanesi-oncology ( Site 1811), Stanbul, Istanbul
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 1801), Ankara
  - Gazi Universitesi-Oncology ( Site 1804), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 1800), Ankara
  - Izmir Atatürk Training and Research Hospital ( Site 1810), Izmir
  - Memorial Kayseri Hastanesi ( Site 1805), Kayseri
  - Mersin Sehir Eğitim ve Araştırma Hastanesi-Oncology ( Site 1808), Mersin
  - Samsun Medical Park Hastanesi-medical oncology ( Site 1806), Samsun
- United Arab Emirates (2):
  - Cleveland Clinic Abu Dhabi ( Site 2650), Abu Dhabi, Abu Dhabi Emirate
  - Burjeel Medical City ( Site 2600), Abu Dhabi, Abu Dhabi Emirate
- United Kingdom (4):
  - North West Cancer Centre ( Site 1908), Londonderry, Derry and Strabane
  - Torbay Hospital ( Site 1906), Torquay, Devon
  - St Bartholomew's Hospital ( Site 1901), London, London, City of
  - City Hospital, Nottingham University Hospitals NHS Trust-NCCTT ( Site 1911), Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26321&tenant=MT_MSD_9011